CLINICAL TRIAL: NCT06401096
Title: Evaluation of the Effects of Preoperative Breathing Exercises on ORI (Oxygen Reserve Index) and ETO2 in Patients Undergoing Abdominal Surgery
Brief Title: Evaluation of the Effects of Preoperative Breathing Exercises on Preoxygenation Period
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, furkan güneş, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-23-4220
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Pre-operative Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control (C): Patients in the control group who will undergo abdominal surgery will not be given any breathing exercises other than routine preoperative preparation. After appropriate anesthesia preparation, preoxygenation will begin.
- Triflo (T): The patient group who receives breathing exercises will be given effective triflo exercise under the supervision of a nurse, starting with hospitalization at least 5 days before the operation and until the pre-operative period. Triflo working time will be planned to be minimum 5 minutes 4 times a day. Breathing exercise will be performed with both inhalation and exhalation. After appropriate anesthesia preparation, preoxygenation will begin.
  Interventions: Procedure: Preoperative respiratory exercises

INTERVENTIONS:
Procedure: Preoperative respiratory exercises — The Triflo Exerciser
  Other Names: Incentive spirometer
  Groups: Triflo (T)

SUMMARY:
The aim of this observational study is to compare the effects of preoperative breathing exercises during the preoxygenation period in patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
Patients who are planned for abdominal surgery under elective conditions and who meet the inclusion criteria will be divided into 2 groups after routine preoperative preparations. The 1st group will start at least 5 days before the preoperative period and until the preoperative period, a minimum of 5 minutes of effective triflo exercise will be performed 4 times a day under the supervision of a nurse, and the 2nd group (control group) will not be exercised except for routine preoperative preparation. Age, existing chronic diseases, body mass index, haemoglobin levels, smoking status, presence or absence of lung disease, SpO2 values before and at the end of respiratory exercise (in the preoperative respiratory exercise group) will be recorded. All patients will be monitored with ECG, SpO2, non invasive blood pressure, Masimo. After the patients are taken to the operating table, they will be preoxygenated with oxygen at FiO2 100% at 10 L\min in supine position, with the anaesthesia mask placed on the patient's face so that there is no leakage. Patients will be preoxygenated until ETO2 concentration reaches 85%. When preoxygenation is started, the timer will be started and the time to reach ORI:0.55 and the time to reach ETO2 85% will be measured and recorded with a timer. Preoxygenation time will be limited to a maximum of 5 minutes and patients who do not reach ETO2 concentration 85% or ORI:0.55 within 5 minutes will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective abdominal surgery under general anesthesia
* Between the ages of 18-65
* Both genders
* ASA I-III risk group
* Patients who accept and give consent to participate in the study

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients younger than 18 years old and older than 65 years old
* Patients with advanced heart failure
* Conditions where the patient is uncooperative (e.g. dementia, Alzheimer's)
* Patients who refuse to breathe through the mask before EtO2 reaches 85% or more after the preoxygenation process begins
* Patients who cannot reach the EtO2 level of 85% within five minutes
* Deeply Anemic Patients (Hb<8 gr/dl)
* Patients with neurological sequelae
* Patients with conditions that may prevent effective preoxygenation (those with long beards, patients with a nasogastric tube, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective abdominal surgery under general anesthesia in Ankara Bilkent City Hospital Operating Room, between the ages of 18-65, both genders and ASA I-III risk group who agree to participate in the study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Duration (sec) for end-tidal oxygen level to rise to 85% | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T)
Duration (sec) for oxygen reserve index to rise to 0.55 | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T)

SECONDARY OUTCOMES:
Duration (sec) for end-tidal oxygen level to rise to 85% according to patient's age | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) according to patient's age
Duration (sec) for oxygen reserve index to rise to 0.55 according to patient's age | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) according to patient's age
Duration (sec) for end-tidal oxygen level to rise to 85% according to patient's BMI | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) according to patient's BMI
Duration (sec) for oxygen reserve index to rise to 0.55 according to patient's BMI | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) according to patient's BMI
Duration (sec) for end-tidal oxygen level to rise to 85% according to patient's gender | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) according to patient's gender
Duration (sec) for oxygen reserve index to rise to 0.55 according to patient's gender | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) according to patient's gender
Duration (sec) for end-tidal oxygen level to rise to 85% depending on whether the patients had known lung disease or not. | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) depending on whether the patients had known lung disease or not.
Duration (sec) for oxygen reserve index to rise to 0.55 depending on whether the patients had known lung disease or not. | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) depending on whether the patients had known lung disease or not.
Duration (sec) for end-tidal oxygen level to rise to 85% according to patient's hemoglobin level | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) according to patient's hemoglobin level
Duration (sec) for oxygen reserve index to rise to 0.55 according to patient's hemoglobin level | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) according to patient's hemoglobin level
Duration (sec) for the end-tidal oxygen level to rise to 85% according to whether the patient smokes or not | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for end-tidal oxygen level to rise 85% of two groups (C and T) according to whether the patient smoked or not.
Duration (sec) for the oxygen reserve index to rise to 0.55 according to whether the patient smokes or not | Between 0th minute and 5th minute of preoxygenation period
  The investigators aimed to compare the duration for oxygen reserve index to rise to 0.55 of two groups (C and T) according to whether the patient smoked or not.
Oxygen saturation level (%) at the beginning and end of 5-day triflo exercise | In the preoperative period before the initiation of triflo exercise and before preoxygenation after 5 days of triflo exercise
  The investigators aimed to examine whether there was a significant difference between oxygen saturations before the start of the study and at the end of the 5-day study in the group of patients who underwent Triflo exercise (T).

CONTACTS AND LOCATIONS:
Overall Officials: Nermin Gögüş, Principal Investigator — Ankara Bilkent City Hospital, Anesthesiology and Reanimation Clinic
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Background] Hulzebos EH, Helders PJ, Favie NJ, De Bie RA, Brutel de la Riviere A, Van Meeteren NL. Preoperative intensive inspiratory muscle training to prevent postoperative pulmonary complications in high-risk patients undergoing CABG surgery: a randomized clinical trial. JAMA. 2006 Oct 18;296(15):1851-7. doi: 10.1001/jama.296.15.1851. PMID 17047215
- [Background] Kundra P, Vitheeswaran M, Nagappa M, Sistla S. Effect of preoperative and postoperative incentive spirometry on lung functions after laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2010 Jun;20(3):170-2. doi: 10.1097/SLE.0b013e3181db81ce. PMID 20551816
- [Background] Chen ST, Min S. Oxygen reserve index, a new method of monitoring oxygenation status: what do we need to know? Chin Med J (Engl). 2020 Jan 20;133(2):229-234. doi: 10.1097/CM9.0000000000000625. PMID 31904726
- [Background] Scheeren TWL, Belda FJ, Perel A. The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):379-389. doi: 10.1007/s10877-017-0049-4. Epub 2017 Aug 8. PMID 28791567